CLINICAL TRIAL: NCT00311727
Title: Cell-Mediated Immune Responses to Influenza A/H5N1 Vaccine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Purpose: Prevention
Other Study IDs: 05-0006
Record Dates: First submitted 2006-04-05; First posted 2006-04-06 (Estimated); Last update posted 2013-08-16 (Estimated); Status verified 2007-05

CONDITIONS: Influenza
Keywords: Cell-Mediated Immune Responses, Influenza, A/H5N1, Vaccine, sub-study
MeSH Terms: conditions — Influenza, Human

ARMS (1):
- Influenza A/H5N1 (Experimental): 232 subjects receiving Influenza A/H5N1 vaccine.
  Interventions: Biological: Influenza A/H5N1

INTERVENTIONS:
Biological: Influenza A/H5N1 — 232 subjects receive Influenza A/H5N1 vaccine as part of DMID protocols 04-063 and 04-076.

SUMMARY:
This study may determine whether laboratory studies of people's blood cells, who have received vaccines against H5 influenza, or "bird flu," will help to decide if the vaccines are going to be prevent disease effectively. About 232 people, 18 years and older, enrolled in the studies "A Randomized, Double-Blinded, Placebo-Controlled, Phase I/II, Dose-Ranging Study of the Safety, Reactogenicity, and Immunogenicity of Intramuscular Inactivated Influenza A/H5N1 Vaccine in Healthy Adults" and "in Healthy Elderly Adults" will participate. Participants may be involved in this study for about 14 months. Procedures may include blood draws, physical exams, and medical history reviews.

DETAILED DESCRIPTION:
This study is linked to DMID protocol 04-063 and 04-076, "A Randomized, Double Blinded, Placebo-ontrolled, Phase I/II, Dose-Ranging Study of the Safety, Reactogenicity, and Immunogenicity of Intramuscular Inactivated Influenza A/H5N1 Vaccine in Healthy Adults (04-063)" and also "in Healthy Elderly Adults" (04-076). All adult subjects enrolled in the main vaccine trials at Vanderbilt (04-076), Maryland (04-063), and Rochester (04-063) will be eligible for enrollment in the cell-mediated immune response sub-study. A maximum of 232 healthy ambulatory male and female subjects; 180 subjects 18 to 64 years old and 64 subjects aged 65 years and older, in the United States, could be enrolled. The primary objectives are: to establish a reproducible, functional cell-mediated immune response assay to evaluate the magnitude and functional capacity of T cells responding to monovalent subvirion H5 influenza vaccine and to evaluate the percent of subjects demonstrating a CD4+ and/or CD8+ response approximately 14 days after the first vaccination and 14 days and 6 months after the second vaccination (04-063), and 14 days after the first and second vaccination and 14 days and 6 months after the third vaccination (04-076). The secondary objectives are: to evaluate dose-related and age-related humoral immunogenicity compared to the cellular immune responses approximately 14 days after the first vaccination and 14 days and 6 months after the second vaccination (04-063), and 14 days after the first and second vaccination and 14 days and 6 months after the third vaccination (04-076) and to establish CMI assays that can be applied to future avian vaccine immunogenicity evaluation, such as the Chiron H9N2 avian influenza vaccine, future H7 vaccines, or vaccines with other avian HA molecules. The study outcome measure, immunogenicity will be based on H5 strain-specific cell-mediated immunity measured 14 days after the first, second, and third (04-076 only) dose, and month 6 after the last dose of vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. All subjects who are eligible and enrolled in the main monovalent subvirion H5 vaccine trials [Division of Microbiology and Infectious Diseases (DMID) studies 04-063 and 04-076] and have agreed to the extra blood draws for the cell-mediated immunity (CMI) sub-study will be enrolled.
2. Subjects will not be recruited outside the main vaccine trials or future DMID sponsored influenza A/H5N1 studies.
3. Subjects who understand and sign the consent form for this study.
4. Subjects who meet pre-screening qualifications for the DMID study will be eligible for the initial pre-vaccination blood draw.
5. Subjects who meet all inclusion criteria for the DMID study and who are vaccinated will be allowed to participate in the remaining portions of this study.

Exclusion Criteria:

1. All subjects who are ineligible for the main monovalent subvirion H5 vaccine trials will not be eligible for the cell-mediated immunity (CMI) sub-study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 339 (Actual)
Dates: Start 2005-10; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Maryland Baltimore, Baltimore, Maryland
  - University of Rochester, Rochester, New York
  - Vanderbilt University, Nashville, Tennessee